CLINICAL TRIAL: NCT03695718
Title: Post-resuscitation Care Registry for Survival From Out-of-hospital Cardiac Arrest
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other); SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jong Hwan Shin, Professor, Seoul National University Hospital
Other Study IDs: 16-2013-157
Record Dates: First submitted 2018-06-08; First posted 2018-10-04 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Out-Of-Hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to construct multi-center post-cardiac arrest care registry that can be used for data warehousing and clinical research.

DETAILED DESCRIPTION:
This registry prospectively enrolls adults patients survived out-of-hospital cardiac arrest in 3 academic hospital emergency departments.

Registered data can be used for quality control and clinical research to reduce post-cardiac arrest syndrome-related mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20 years old or older who presents to the ED of the participating hospitals with any of the following criteria:

  1. Sustained ROSC from OHCA at pre-hospital level
  2. Sustained ROSC from OHCA at the ED of the participating hospitals after ACLS
  3. Patients sustained ROSC from OHCA and transferred from other hospital to the ED of the participating hospitals for post-cardiac arrest care

Exclusion Criteria:

* Age less than 20 years old
* Patients with advanced directives not to deliver aggressive organ supportive management

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with sustained ROSC from OHCA
Sampling Method: Non-Probability Sample
Enrollment: 1057 (Actual)
Dates: Start 2013-12-03 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Survival | 1-year
  One year survival

SECONDARY OUTCOMES:
28-day mortality | 28-day
  Mortality on the 28th day
28-day CPC | 28-day
  Brain function at 28th day
6-month CPC | 6-month
  Brain function at 6-month
1-year CPC | 1-year
  Brain function at 1-year
Organ support treatment (mechanical ventilation) | Hospital discharge (non-survivors) or 1-year (survivors)
  Mechanical ventilation
Organ support treatment (renal replacement therapy) | Hospital discharge (non-survivors) or 1-year (survivors)
  Renal replacement therapy
ICU length of stay | Hospital discharge (non-survivors) or 1-year (survivors)
  ICU length of stay
Hospital length of stay | Hospital discharge (non-survivors) or 1-year (survivors)
  Hospital length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Jonghwan Shin, MD, PhD, Study Director — Seoul National University Boramae Hospital
Locations (3):
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Seoul National University Boramae Hospital, Seoul